CLINICAL TRIAL: NCT00793065
Title: Evaluating the Effects of EHRs, P4P and Medical Home Redesign in the Hudson Valley
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York State Department of Health (Other Government); The Commonwealth Fund (Other); Taconic Health Information Network and Community (THINC) (Unknown); Taconic Independent Practice Association (TIPA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0508190240
Record Dates: First submitted 2008-11-14; First posted 2008-11-19 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Quality of Health Care; Electronic Health Records
Keywords: electronic health records; health information technology; physician incentives; quality of health care
MeSH Terms: interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Physicians that are using paper-based medical charts and who are not receiving Medical Home redesign incentives.
- 2: Physicians that are using Electronic Health Records (EHRs) and who are not undergoing Medical Home redesign.
  Interventions: Other: Electronic health record (EHR)
- 3: Physicians that are using Electronic Health Records (EHRs) and undergoing Medical Home redesign.
  Interventions: Other: Electronic health record (EHR); Other: Medical Home redesign

INTERVENTIONS:
Other: Electronic health record (EHR) — Computer-based system that allows physicians to access and manage patient records electronically.
  Groups: 2; 3
Other: Medical Home redesign — Implementation of NCQA Level III Medical Home
  Groups: 3

SUMMARY:
The investigators will conduct a longitudinal cohort study with concurrent controls. The investigators will include all primary care physicians in the Hudson Valley including family practitioners, internists, and pediatricians. The purpose of this study is to determine the effects of implementing electronic health records (EHRs), pay-for-performance incentives for physicians (P4P), and Medical Home redesign on health care quality, cost and patient experience in the Hudson Valley.

DETAILED DESCRIPTION:
The Hudson Valley is implementing several innovative programs to potentially improve quality and reduce the cost of health care delivered. First the Taconic Health Information Network and Communities Regional Health Information Organization (THINC RHIO) is facilitating diffusion of EHRs in office practices in the Hudson Valley. Second, THINC RHIO is also offering a strategic approach to pay-for-performance. Third, an additional component of the THINC P4P project will be an added financial incentive for private practice physicians who implement and reach Level II of Physician Practice Connections® - Patient Centered Medical Home (PCMH)™, NCQA's new national recognition system for physician practices. Our study will seek to determine the effect of each of these initiatives on health care quality and cost of care in the Hudson Valley. We will also measure the patient experience before and after implementation of the Medical Home.

ELIGIBILITY:
Inclusion Criteria:

* Primary care physicians working in the offices practices in the Hudson Valley, and who are members of the Taconic IPA.

Exclusion Criteria:

* Physicians who opt out from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All primary care physicians (i.e. general internists, pediatricians and family practice physicians) in the Hudson Valley who are members of the Taconic Independent Practice Association (IPA).
Sampling Method: Non-Probability Sample
Enrollment: 438 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
health care quality (as determined by previously selected and approved quality indicators) | 5 years
health care utilization | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Kern, MD, MPH, Principal Investigator — Weill Medical College of Cornell University; Rainu Kaushal, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Derived] Kern LM, Edwards A, Kaushal R. The Patient-Centered Medical Home and Associations With Health Care Quality and Utilization: A 5-Year Cohort Study. Ann Intern Med. 2016 Mar 15;164(6):395-405. doi: 10.7326/M14-2633. Epub 2016 Feb 16. PMID 26882534
- [Derived] Kaushal R, Edwards A, Kern LM; HITEC Investigators. Association between electronic health records and health care utilization. Appl Clin Inform. 2015 Jan 28;6(1):42-55. doi: 10.4338/ACI-2014-10-RA-0089. eCollection 2015. PMID 25848412
- [Derived] Kern LM, Edwards A, Kaushal R. The patient-centered medical home, electronic health records, and quality of care. Ann Intern Med. 2014 Jun 3;160(11):741-9. doi: 10.7326/M13-1798. PMID 24887615